CLINICAL TRIAL: NCT06029036
Title: A Phase II, Multi-center, Single-arm, Prospective Study of Darolutamide + ADT Prior to Radical Prostatectomy (RP) in High-risk/Very High-risk Localized Prostate Cancer
Brief Title: A Phase II Neoadjuvant Study of Darolutamide Plus ADT in Men With Localized Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22440
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Darolutamide + ADT (Experimental): Duration of treatment: 28-day cycle of darolutamide treatment and 6 cycles of neoadjuvant therapy.
  Interventions: Drug: Darolutamide+ADT

INTERVENTIONS:
Drug: Darolutamide+ADT — Drug: Darolutamide
  Darolutamide 600 mg, (two 300 mg tablets) administered orally twice daily. Swallow tablets whole. Take Darolutamide with food.
  Drug: ADT GnRH agonist per physicians' choice, orchiectomy is excluded

SUMMARY:
Scientific Rationale: High risk localized prostate cancer (PCa) is associated with higher rates of biochemical recurrence, clinical recurrence, metastasis and PCa-specific death. Novel hormone therapies(NHT) have shown a significant survival advantage with respect to classical ADT in later stages of PCa and have already been investigated in neoadjuvant setting.

PURPOSE: To assess antitumor effect by measuring pathological tumor volume with pathological downstaging following radical prostatectomy + pelvic lymph-node dissection (RP + PLND) for high-risk localized prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥18 years of age.
2. Able to Sign informed consent form independently.
3. Non-metastatic adenocarcinoma of the prostate.
4. Subjects must have as least one of the following features according to NCCN definition of high-risk: Gleason score ≥8, or PSA >20ng/ml,or≥clinical T3a.
5. Subjects with pelvic lymph node involvement(N1) can be included.
6. Candidate for radical prostatectomy with or without pelvic lymph node dissection as per the investigator.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
8. Subjects must have normal organ and marrow function as defined below:

Hemoglobin ≥ 9.0 g/dL;Absolute neutrophil count (ANC) ≥ 1,500/mcL; Platelets ≥ 100,000/mcL, independent of transfusions/growth factors within 3 months of treatment start; Serum potassium ≥ 3.5 mmol/L; Serum total bilirubin ≤ 2.0 x upper limit of normal (ULN) (except in subjects with Gilbert's syndrome who have a total bilirubin > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1.5 x ULN, subject may be eligible);Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN;Serum albumin ≥ 3.0 g/dL;Serum creatinine < 2.0 x ULN.

Exclusion Criteria:

1. Prostate cancer with neuroendocrine differentiation or small cell features
2. Distant metastasis based on conventional imaging (clinical stage M1). Nodal disease below the iliac bifurcation (clinical stage N1) is not an exclusion.
3. History of prior systemic or local therapy for prostate cancer, including pelvic radiation for prostate cancer.
4. Subjects who are planning bilateral orchidectomy during the treatment period of the study.
5. Intolerable with darolutamide or ADT treatment.
6. Candidates of other clinical trials.
7. Any prior malignancy within 5 years.
8. Complications include significant cardiovascular disease, active infection, astrointestinal disorders, or any other complications that in the opinion of the investigator.
9. Any condition that in the opinion of the investigator would preclude participation in this study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological downstaging | 6 months
  Percentage of patients with tumor downstaging

SECONDARY OUTCOMES:
pCR or MRD | 6 months
  Pathologic complete response or Minimal Residual Disease(defined as overall diameter <5 mm)
PSM | 6 months
  Percentage of patients with positive surgical margins
Rate of peri-operative complications | within 30 days of surgery
  including delay in surgery, intra-operative complications, and postoperative complications
Biochemical complete response | 6 months
  PSA <0.1ng/ml prior to RP
PSA undetectable rate | 12 months post-RP
  PSA<0.02 ng/ml
2-year biochemical progression-free survival, bPFS | 24 months post-RP
  PSA>0.2 ng/ml
AEs/SAEs | Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first
  The level of AEs defined by NCI-CTCAE v5.0. Safety assessments will be assessed and documented after initiation of study drug, regardless of relationship to study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No